CLINICAL TRIAL: NCT01061879
Title: Ex Vivo Expansion of Umbilical Cord Blood Using a Unique Bio-system
Brief Title: Expansion of Umbilical Cord Blood Using a Unique Bio-system
Status: Completed | Type: Observational
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 11973
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Pregnancy
Keywords: umbilical cord; umbilical cord blood collection; pregnancy

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — umbilical cord
Oversight: Data Monitoring Committee: No

SUMMARY:
By doing this study, researchers hope to develop a special technique and laboratory conditions to help support umbilical stem cell growth and multiplication.

In this project, researchers propose a three dimensional (3D) microenvironment that mimics the bone marrow stem cell microenvironment, with its supporting cells of osteoblasts and stromal cells. In theory, this will result in better expansion of cord blood stem cells ex vivo.

DETAILED DESCRIPTION:
To successfully expand umbilical cord blood stem cells ex vivo, a microenvironment that resembles the stem cell microenvironment, or stem cell 'niche' should be created. In designing this bio-system, we make use of several observations. First, bone osteoblasts are important in promoting hematopoietic stem cell expansion, accordingly, this bio-system will ensure the physical proximity of the cord blood stem cells to a 3D bone tissue derived from mesenchymal stem cells (MSCs). These MSCs will be isolated from Wharton's jelly, and by using an osteogenic medium and special scaffolds, these MSCs will differentiate into osteogenic progenitors creating a 3D bone structure. The other observation is that, co-culture of cord blood stem cells with mesenchymal stem cells is superior to liquid cultures in terms of ex vivo expansion , accordingly, in this experiment, undifferentiated MSCs will be co-cultured with cord blood stem cells in this created 3D bone structure. This is a unique design that has the potential to expand cord blood stem cells more efficiently.

ELIGIBILITY:
Inclusion Criteria:

* females that consent to permit researchers collect the discarded umbilical cords from the placenta and use for research purposes.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: umbilical cord collection from full-term caesarian section/normal vaginal delivery patients
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
bio-system for ex-vivo expansion of umbilical cord blood stem cells | one year
  To successfully expand the umbilical cord blood stem cells, a microenvironment that resembles the stem cell microenvironment, or stem cell 'niche' should be created. In designing this bio-system, we make use of several observations. Firstly, bone osteoblasts are important in promoting hematopoietic stem cell expansion , accordingly, this bio-system will ensure the physical proximity of the cord blood stem cells to a 3D bone tissue derived from mesenchymal stem cells (MSCs). These MSCs will be isolated from Wharton's jelly, and by using an osteogenic medium and special scaffolds, these MSCs will differentiate into osteogenic progenitors creating a 3D bone structure . The other observation is that, co-culture of cord blood stem cells with mesenchymal stem cells is superior to liquid cultures in terms of ex vivo expansion , accordingly, in this experiment, undifferentiated MSCs will be co-cultured with cord blood stem cells in the created 3D bone structure.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Aljitawi, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States